CLINICAL TRIAL: NCT00066222
Title: A Phase II Study Of Accelerated High Dose Thoracic Irradiation With Concurrent Chemotherapy For Patients With Limited Small Cell Lung Cancer
Brief Title: Cisplatin, Etoposide, and Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0239; CDR0000271939
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Therapy + Chemotherapy (Experimental): Accelerated high dose thoracic radiation therapy (RT) with concurrent cisplatin/etoposide chemotherapy, followed by 2 cycles of adjuvant cisplatin/etoposide chemotherapy
  Interventions: Drug: Cisplatin; Drug: Etoposide; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Cisplatin — 60 mg/m2 given intravenously. During RT, give on day 1 and day 22. After completion of RT, on days 43 and 64.
Drug: Etoposide — 120 mg/m2 given intravenously. During RT, give on days 1-3, then days 22-24. After completion of RT, on days 43-45 and days 64-66.
Radiation: Radiation therapy — Large field 28.8 Gy: 1.8 Gy per fraction, 5 days per week for 16 fractions. On days 23-26, BID: use anteroposterior and posteroanterior (AP/PA) fields in a.m. at 1.8 Gy per fraction; boost with 2nd treatment in p.m. at 1.8 Gy per fraction. Then off-cord boost, 1.8 Gy, BID, x last 5 days for a total dose of 61.2 Gy in 5 wks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin and etoposide together with radiation therapy works in treating patients with limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with limited stage small cell lung cancer treated with cisplatin and etoposide combined with accelerated high-dose thoracic radiotherapy.
* Determine the progression-free and overall survival in patients treated with this regimen.
* Determine the qualitative and quantitative toxicity and reversibility of toxicity of this regimen in these patients.

OUTLINE: Patients undergo radiotherapy once daily 5 days a week for approximately 3 weeks and then twice daily 5 days a week for approximately 2 weeks (a total of 9 treatment days during the final 2-week treatment period). Beginning on the first day of radiotherapy, patients receive cisplatin IV over 2 hours and etoposide IV over 1 hour on day 1 and oral etoposide once daily on days 2 and 3. Chemotherapy repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell carcinoma of the lung by fine needle aspiration biopsy or two positive sputa
* Must have limited disease

  * Stage I, II, IIIA, or IIIB

    * Confined to 1 hemithorax, but excluding the following:

      * T4 tumor based on malignant pleural effusion
      * N3 disease based on contralateral hilar or contralateral supraclavicular involvement
* No pericardial or pleural effusions on chest x-ray (regardless of cytology)
* Measurable or evaluable disease
* Tumor must be able to be encompassed by limited radiotherapy fields without significantly compromising pulmonary function
* No prior complete tumor resection

PATIENT CHARACTERISTICS:

Age

* 18 to 100

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No symptomatic heart disease

Pulmonary

* No chronic obstructive pulmonary disease with Forced Expiratory Volume (FEV)-1 no greater than 0.8 liter
* No uncontrolled bronchospasm in the unaffected lung

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Available for follow-up
* No other malignancy within the past 2 years except curatively treated basal cell or squamous cell skin cancer or non-invasive in situ malignancies
* No other concurrent serious medical illness
* No uncontrolled psychiatric illness
* No chronic alcohol or drug abuse

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the chest or other area containing a large amount of bone marrow (e.g., more than 75% of pelvic bone)

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2003-06; Primary Completion 2012-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritsuko U. Komaki, MD, FACR, Study Chair — M.D. Anderson Cancer Center
Locations (104):
- United States (104):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - Eden Medical Center, Castro Valley, California
  - Saint Rose Hospital, Hayward, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Robert and Beverly Lewis Family Cancer Care Center at Pomona Valley Hospital Medical Center, Pomona, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Wendt Regional Cancer Center at Finley Hospital, Dubuque, Iowa
  - Cancer Treatment Center at the Medical Center - Bowling Green, Bowling Green, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - St. Agnes Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Fox Chase Cancer Center at St. Francis Medical Center, Trenton, New Jersey
  - South Jersey Healthcare Regional Cancer Center, Vineland, New Jersey
  - Fitzpatrick Cancer Center at Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Wilmed Radiation Oncology Services, Wilson, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Huron Hospital Cancer Care Center, Cleveland, Ohio
  - Euclid Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Cancer Research UK Medical Oncology Unit at Churchill Hospital & Weatherall Institute of Molecular Medicine - Oxford, Salem, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital Cancer Care Center, Warrensville Heights, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Columbia St. Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Result] Komaki R, Paulus R, Ettinger DS, Videtic GM, Bradley JD, Glisson BS, Langer CJ, Sause WT, Curran WJ Jr, Choy H. Phase II study of accelerated high-dose radiotherapy with concurrent chemotherapy for patients with limited small-cell lung cancer: Radiation Therapy Oncology Group protocol 0239. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):e531-6. doi: 10.1016/j.ijrobp.2012.01.075. Epub 2012 May 5. PMID 22560543
- [Result] Komaki R, Paulus R, Ettinger DS, et al.: A phase II study of accelerated high-dose thoracic radiation therapy (AHTRT) with concurrent chemotherapy for limited small cell lung cancer: RTOG 0239. [Abstract] J Clin Oncol 27 (Suppl 15): A-7527, 2009.
- [Result] Komaki R, Moughan J, Ettinger D, et al.: Toxicities in a phase II study of accelerated high dose thoracic radiation therapy (TRT) with concurrent chemotherapy for limited small cell lung cancer (LSCLC) (RTOG 0239). [Abstract] J Clin Oncol 25 (Suppl 18): A-7717, 438s, 2007.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy + Chemotherapy
Started | 72
Completed | 71 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 1
Not completed — No protocol treatment received | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who started protocol treatment.
Groups:
- Radiation Therapy + Chemotherapy: Accelerated high dose thoracic RT with concurrent cisplatin/etoposide chemotherapy, followed by 2 cycles of adjuvant cisplatin/etoposide chemotherapy
Arm/Group | Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 71
Age, Continuous [Median (Full Range); unit: years] | 71 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 2 Years
Description: Survival time is defined as time from study registration to the date of death from any cause and survival rates are estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From registration to 2 years
Population: All eligible patients who started study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 71
percentage of participants | 36.60 [25.60 to 47.70]
Statistical Analysis 1: Comparison: Radiation Therapy + Chemotherapy; This study was designed to detect an improvement in the 2-year overall survival rate from 47% to 60%. Using a one-group chi-square test with a one-sided significance level of 0.10, a sample of 67 patients was deemed sufficient to detect the difference between the null hypothesis (H0: P .47) and the alternative hypothesis (HA: P .60) with 80% power; Test type: Other; If the point estimate for two-year survival is less than or equal to 0.54815, the upper bound of the one-sided 90% confidence interval on 47%, then H0 would not be rejected and the conclusion would be that the two-year survival rate did not statistically improve from 47% under the new treatment. If the point estimate is greater than 0.54815, then H0 would be rejected and the conclusion is that the two-year survival rate did improve from 47% to 60% under the new treatment

2. Secondary Outcome: Overall Survival (OS) and Progression-free Survival (PFS) at 1 Year
Description: An event for overall survival is death due to any cause. Overall survival time is defined as time from study registration to the date of death from any cause. An event for progression-free survival is the first of the following: local progression, regional progression, distant metastases, or death due to any cause. Progression-free survival time is defined as time from study registration to the date of first failure. For both outcome measures, patients last known to be alive without failure are censored at the date of last contact. Survival rates are estimated by the Kaplan-Meier method.
Time Frame: From registration to one year.
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 71
percentage of participants
  Overall Survival | 77.5 [65.9 to 85.5]
  Progression-free Survival | 42.3 [30.7 to 53.4]

3. Secondary Outcome: Median Overall Survival Time and Progression-free Survival Time
Description: as for outcome 2
Time Frame: From registration to 2 years
Population: All eligible patients who started study treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 71
months
  Overall Survival | 19.0 [16.7 to 21.7]
  Progression-free Survival | 9.9 [7.9 to 12.4]

4. Secondary Outcome: Number of Patients With Acute Treatment-related Grade 3 or 4 Esophagitis
Description: Highest grade treatment-related toxicity per subject was counted. Toxicities were graded using Common Toxicity Criteria (CTC) v 2.0. Grade refers to the severity of the toxicity. Both criteria assign Grades 1 through 5 with unique clinical descriptions of severity for a given toxicity based on this general guideline: Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening or disabling, Grade 5= Death related to toxicity.
Time Frame: From start of radiation therapy until 90 days following the start of radiation therapy
Population: Eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 71
Participants | 13
Statistical Analysis 1: Comparison: Radiation Therapy + Chemotherapy; Test type: Other; The following rule would reject the null hypothesis that the proportion of severe esophagitis was 30% with an overall significance level of 0.05: 27 or more cases of severe esophagitis among the total sample of evaluable patients

5. Secondary Outcome: Frequency of Treatment-related Fatalities at 2 Years
Description: A treatment-related fatality was any death judged to be related to protocol treatment.
Time Frame: From the start of treatment to 2 years
Population: Eligible patients who started study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 71
Participants | 2
Statistical Analysis 1: Comparison: Radiation Therapy + Chemotherapy; Test type: Other; The following rule would reject the null hypothesis that the proportion of treatment-related fatalities was less than or equal to 5% with an overall significance level of 0.05: 6 or more instances of treatment-related fatalities among the total sample of evaluable patients

6. Secondary Outcome: Tumor Response
Description: Response will be recorded as the best response observed two months after the completion of chemoradiation therapy. Tumor response as defined by Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR): Disappearance of all target lesions as measured by MRI, CT, or physical examination (this is the order of preference for measurement). Partial Response (PR): >= 30% decrease in the sum of the longest diameter (LD) of target lesions (order of preference for measurement is MRI, CT, physical examination). Progressive Disease (PD): >= 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions (order of preference for measurement is MRI, CT, physical examination). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: From the start of treatment to 2 months following the completion of chemotherapy
Population: Eligible patients who started study treatment and were observed for at least 2 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 68
Participants
  Complete Response | 29
  Partial Response | 28
  Stable Disease | 7
  Progressive Disease | 4

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events (AE).
Arm/Group | Radiation Therapy + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 67/71
Other Adverse Events (participants affected / at risk) | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy + Chemotherapy (N=71)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 14
Hematologic-Other (Blood and lymphatic system disorders) | 1
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 18
Hemoglobin (Hgb) for leukemia (Blood and lymphatic system disorders) | 1
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis, other) (Blood and lymphatic system disorders) | 1
Thrombotic microangiopathy for BMT (e.g., thrombotic thrombocytopenic purpura/TTP or hemolytic urem (Blood and lymphatic system disorders) | 1
Transfusion: Platelets (Blood and lymphatic system disorders) | 2
Transfusion: pRBCs (Blood and lymphatic system disorders) | 2
Arrhythmia- other (Cardiac disorders) | 1
Circulatory or cardiac-Other (Cardiac disorders) | 1
Late RT Toxicity: Heart: NOS (Cardiac disorders) | 1
Pericardial effusion/pericarditis (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (without colostomy) (Gastrointestinal disorders) | 2
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 7
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 6
GI-Other (Gastrointestinal disorders) | 1
Mucositis due to radiation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 12
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 109/L) (General disorders) | 1
Pain-Other (General disorders) | 4
Hepatic-Other (Hepatobiliary disorders) | 1
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 7
Infection with unknown ANC (Infections and infestations) | 1
Infection without neutropenia (Infections and infestations) | 3
Infection, Other (Infections and infestations) | 1
Wound-infectious (Infections and infestations) | 1
Operative injury of vein/artery (Injury, poisoning and procedural complications) | 1
Bilirubin (Investigations) | 1
Cardiac troponin T (cTnT) (Investigations) | 1
Creatinine (Investigations) | 3
Leukocytes (total WBC) (Investigations) | 53
Lymphopenia (Investigations) | 7
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 56
Platelets (Investigations) | 4
SIADH (syndrome of inappropriate anti-diuretic hormone) (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesmia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 9
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Memory loss (Nervous system disorders) | 1
Neuropathic pain (e.g., jaw pain, neurologic pain, phantom limb pain, post-infectious neuralgia, or (Nervous system disorders) | 3
Neuropathy motor (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 2
Seizure(s) (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 4
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Late RT Toxicity: Lung: NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 3
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Peripheral arterial ischemia (Vascular disorders) | 1
Thrombosis/embolism (Vascular disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy + Chemotherapy (N=71)
Hematologic-Other (Blood and lymphatic system disorders) | 5
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 48
Edema (Cardiac disorders) | 5
Constipation (Gastrointestinal disorders) | 17
Diarrhea (without colostomy) (Gastrointestinal disorders) | 11
Dyspepsia/heartburn (Gastrointestinal disorders) | 6
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 25
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 24
Dysphagia-pharyngeal related to radiation (Gastrointestinal disorders) | 4
GI-Other (Gastrointestinal disorders) | 6
Late RT Toxicity: Esophagus: NOS (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 38
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 24
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 5
Fatigue (lethargy, malaise, asthenia) (General disorders) | 55
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 109/L) (General disorders) | 6
Late RT Toxicity: Other: NOS (General disorders) | 17
Pain due to radiation (General disorders) | 9
Pain-Other (General disorders) | 11
Late RT Toxicity: Skin: NOS (Injury, poisoning and procedural complications) | 7
Radiation dermatitis (Injury, poisoning and procedural complications) | 18
Alkaline phosphatase (Investigations) | 4
Creatinine (Investigations) | 14
Leukocytes (total WBC) (Investigations) | 10
Lymphopenia (Investigations) | 7
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 6
Platelets (Investigations) | 48
Weight loss (Investigations) | 20
Anorexia (Metabolism and nutrition disorders) | 33
Dehydration (Metabolism and nutrition disorders) | 19
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesmia (Metabolism and nutrition disorders) | 17
Hyponatremia (Metabolism and nutrition disorders) | 13
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 6
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 4
Ataxia (incoordination) (Nervous system disorders) | 5
Dizziness/lightheadedness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 8
Memory loss (Nervous system disorders) | 5
Neuropathy motor (Nervous system disorders) | 4
Neuropathy-sensory (Nervous system disorders) | 7
Taste disturbance (dysgeusia) (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 6
Mood alteration-depression (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 17
Late RT Toxicity: Lung: NOS (Respiratory, thoracic and mediastinal disorders) | 37
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 30
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.